CLINICAL TRIAL: NCT03903497
Title: Efficacy of WASP Classification in the Histological Evaluation of Diminutive Colorectal Polyps
Brief Title: WASP Classification in Diagnosis of Diminutive Colorectal Polyps
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Beijing Friendship Hospital (Other); Jilin People's Hospital (Unknown); Wafangdian Third Hospital (Unknown); Dezhou People's Hospital (Other); Liaocheng People's Hospital (Other); Wenzhou Central Hospital (Other); Yichun People's Hospital (Unknown); The Third Xiangya Hospital of Central South University (Other); Shenzhen Baoan People's Hospital (Unknown); Xinxiang Central Hospital (Other); Wuwei Cancer Hospital (Unknown); Zunyi Medical College (Other); Yaan People's Hospital (Unknown)
Responsible Party: Principal Investigator, Zhizheng Ge, MD,Ph.D, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: rj[2018]086
Record Dates: First submitted 2019-04-01; First posted 2019-04-04 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Diminutive Colorectal Polyps
Keywords: Narrow band imaging; WASP classification; Diminutive colorectal polyps

STUDY DESIGN:
Intervention Model Description: Colonoscopy with NBI using the WASP classification
Masking Description: Endoscopists did not know histology of diminutive colorectal polyps
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NBI assessment using the WASP classification (Other)
  Interventions: Device: NBI

INTERVENTIONS:
Device: NBI — optical assessment of diminutive colorectal polyps by NBI mode using the WASP assessment

SUMMARY:
Adenomas, serrated adenomas and hyperplastic polyps are polypoid lesion in the colorectum. At the present moment, all polyps should be resected endoscopically, although only adenomas and serrated adenomas, but not hyperplastic polyps have the potential to develop colorectal cancer. Some studies have investigated the value of the narrow-band imaging (NBI) on histological prediction of the polyp. This method is conducted in real time during colonoscopy, which leads to simplification of diagnostic procedures. For instance, it would be conceivable to resect diminutive polyps and discard them without further assessment by a pathologist. One problem in this context is a correct differentiation between hyperplastic polyps and serrated adenomas. These two polyp entities are known to show similar optical features. However, while serrated adenomas are premalignant lesions hyperplastic polyps have benign histology and never develop into cancer. It is therefore important to sufficiently distinguish hyperplastic polyps from serrated lesions.

In this study the investigators want to investigate whether the use of NBI would be capable to get accuracy of optical polyp predictions by more than 90% using the WASP (Workgroup serrAted polypS and Polyposis) classification. NBI is a light filter tool which can be activated by pressing a button at the endoscope. The use of NBI leads to an endoscopic picture which appears blue and enables endoscopists to better assess surface structures and vascular patterns. All polyps will be resected and send to pathology for further microscopic assessment. After completing the trial the investigators aim to compare accuracy of the optical diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged more than 18 years old
* Patients with at least one diminutive colorectal polyp

Exclusion Criteria:

* Patients with poor bowel preparation
* Paitents with history of colorectal surgery, familial adenomatous polyposis or inflammatory bowel disease
* Patients with advanced colorectal cancer
* Patients with missed histology information of resected polyps or missed resected specimen
* Patients with emergency operation during colonoscopy
* Patients with unfinished colonoscopy due to any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2640 (Estimated)
Dates: Start 2019-04-15 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
Accuracy of Surveillance time prediction of patients with at least one diminutive polyps under high confidence of diagnosis | Within two weeks after polypectomy
Negative predictive value of diminutive polyps located in rectum and sigmoid colon under high confidence of diagnosis | Within two weeks after polypectomy
Accuracy of WASP classification in histological prediction of diminutive polyps under high confidence of diagnosis | Within two weeks after polypectomy

SECONDARY OUTCOMES:
Learning curve of accuracy of endoscopists using NBI in assessment of diminutive polyps | Within two weeks after polypectomy

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing Friendship Hospital, Beijing, Beijing Municipality
  - Renji Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No